CLINICAL TRIAL: NCT05185609
Title: Assessment of Anorectal Function in Healthy Volunteers and Patients With Inflammatory Bowel Disease
Brief Title: Assessment of Anorectal Function in Patients With Inflammatory Bowel Disease
Status: Recruiting | Type: Observational
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Other Study IDs: Regionorebrolan 252641
Record Dates: First submitted 2021-11-24; First posted 2022-01-11 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2021-12

CONDITIONS: Inflammatory Bowel Diseases; Irritable Bowel Syndrome
Keywords: Anorectal function; Anorectal manometry; Rectal barostat
MeSH Terms: conditions — Inflammatory Bowel Diseases; Irritable Bowel Syndrome | interventions — Compliance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Serum. Stool samples. Rectal mucosal biopsies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy volunteers: Healthy volunteers aged 18-to 65
  Interventions: Other: Exposure 1: Visceral hypersensitivity or phenotype suggestive of IBS; Other: Exposure 2: Changes in anorectal motor function or compliance.
- Asymptomatic patients with quiescent IBD: Asymptomatic patients with IBD in remission.
  Interventions: Other: Exposure 1: Visceral hypersensitivity or phenotype suggestive of IBS; Other: Exposure 2: Changes in anorectal motor function or compliance.
- Symptomatic patients with quiescent UC: Symptomatic patients with UC in remission
  Interventions: Other: Exposure 1: Visceral hypersensitivity or phenotype suggestive of IBS; Other: Exposure 2: Changes in anorectal motor function or compliance.
- Symptomatic patients with quiescent CD with anorectal involvement: Symptomatic patients with CD with distal involvement of the colon or perianal disease
  Interventions: Other: Exposure 1: Visceral hypersensitivity or phenotype suggestive of IBS; Other: Exposure 2: Changes in anorectal motor function or compliance.

INTERVENTIONS:
Other: Exposure 1: Visceral hypersensitivity or phenotype suggestive of IBS — Assess the relation between the exposure and the outcome which is persistent symptoms in the patients with quiescent disease.
Other: Exposure 2: Changes in anorectal motor function or compliance. — Assess the relation between the exposure and the outcome which is persistent symptoms in the patients with quiescent disease.

SUMMARY:
Active inflammatory bowel disease (IBD) causes disabling symptoms such as diarrhea, involuntary loss of bowel control, abdominal pain and urges to pass stool. However, even patients with inactive IBD frequently experience such symptoms. The cause is not well understood and the functionality of the bowel in IBD patients is underexplored.

Earlier studies show a wide range of results, but most find that patients with IBD in remission are up to four times as likely to report gastrointestinal symptoms when compared to healthy controls.

Chronic inflammation may cause changes of the bowel wall, like increased collagen deposits (fibrosis) and thus cause symptoms, but the absence of active inflammation in combination with presence of symptoms may also be regarded as resembling the clinical condition of irritable bowel syndrome (IBS).

IBS is characterized by abdominal pain and changes in stool frequency and consistence and is often associated with disorders like depression and anxiety. Up to a third of IBD patients without signs of disease activity meet the criteria for IBS (irritable bowel syndrome. It can be speculated that an IBD diagnosis is a distressing event that can induce mood disorders, and an IBS-like condition.

Characterization of IBS patients relies on the Rome IV symptom criteria, symptom severity scales and measurements of rectal sensibility and rectal compliance using a barostat procedure.

Motor function assessment relies on anorectal manometry which detects abnormalities of muscle function and coordination. Recently, a standardized high-resolution anorectal manometry protocol (HRAM) was published which also evaluates sensitivity and compliance. The level of agreement between the barostat method and the HRAM testing procedure regarding sensibility and rectal compliance is largely unknown.

Recent studies have associated gut microorganisms, genetic factors, and proteins with various aspects of IBD. There is evidence that these potential markers may reflect non-inflammatory processes such as fibrosis.

The aim of this study is to explore the anorectal function in symptomatic patients with inactive IBD compared to healthy volunteers and asymptomatic patients, evaluate symptom severity and psychological parameters and perform molecular characterization.

The level of agreement of rectal sensitivity and compliance measurements with the barostat method and HRAM protocol will also be evaluated.

DETAILED DESCRIPTION:
Anorectal function (ARF) disorders in patients with IBD cause disabling symptoms such as fecal incontinence, increases in the stool frequency, urgency and tenesmus.

Patients with IBD in remission frequently experience diarrhea, fecal incontinence and lower GI symptoms. However, ARF in IBD patients is underexplored.

Chronic mucosal inflammation may induce visceral hypersensitivity and rectal wall fibrosis, but the casual relationship is hypothetical.

The absence of active inflammation and the presence of symptoms resemble IBS leading to the speculation that an IBD diagnosis is a distressing event, and can induce mood disorders, and an IBS-like condition.

Anorectal manometry detects abnormalities of sphincter function and rectoanal coordination. Recently, a standardized HRAM protocol was published (The London consensus protocol) witch also evaluates rectal sensitivity (RS) and rectal compliance (RC).

Earlier studies, using water-perfused AM, indicated that patients with active ulcerative colitis (UC) may have increased RS, contractility and impaired RC whereas patients with quiescent UC may have impaired RC, suggesting that chronic fibrotic changes of the rectal wall may occur.[14, 15] IBS is characterized by abdominal pain and changes in stool pattern. Its biological hallmark is increased visceral perception with disturbed bidirectional brain-gut signaling, associated with serotonergic dysregulation, illustrated by the high prevalence of mood disorders.

IBS is diagnosed using the Rome IV symptom criteria. Phenotyping IBS patients, as described in a consensus paper by Boeckxstaens et al. in 2017, relies on GI symptom severity scales and measurements of RS and RC using a barostat procedure. There is frequently overlap with other functional GI disorders (FGIDs). Hence these should also be assessed, as well as psychological comorbidities.

The gold standard for phenotyping is the use of validated questionnaires and a standardized barostat protocol as described in a publication from the European COST action GENIEUR group.[16] The level of agreement between the barostat protocol and the HRAM testing procedure regarding sensory testing and measurement of rectal compliance is not established.

Progress in various types of -omics techniques has enhanced our possibilities to identify markers of complex diseases such as IBD. Recent studies have associated gut microbiota, genome, transcriptome and proteome-profiles with various aspects of the disease. Both individual markers and panels of markers, so called "molecular signatures" are currently tested for their predictive capacity and possible source for future biomarker identification. Accumulating data indicate that some of this novel potential markers may reflect non-inflammatory processes such as fibrosis.

The overarching aim of this study is to explore the anorectal function in symptomatic patients with quiescent IBD compared to healthy volunteers and asymptomatic patients with quiescent IBD, using both HRAM and a standardized barostat procedure. Symptom severity and psychological parameters will be evaluated by validated questionnaires. Molecular characterization will be performed by analyses of blood, faecal samples and mucosal biopsies.

Examination of single-layers of molecular data will be followed by integrated analyses of several layers of - omics data and correlated to clinical and psychological phenotypes. This "multi-omics" approach requires development of bioinformatic methods, which currently are underway.

The study goals are:

1. To determine the level of agreement and correlation of rectal sensitivity- and compliance measurements between the HRAM method and the barostat method in healthy volunteers and asymptomatic patients with IBD in remission
2. To study ARF in symptomatic patients with IBD in remission and to compare the results with data from healthy volunteers and asymptomatic patients with IBD in remission.
3. To measure parameters of brain-gut interaction in IBD patients using validated GI symptom scales and psychometric questionnaires on anxiety, somatization, personality and depression and to compare the results with data from healthy volunteers.
4. To analyse plasma, stool and rectal mucosa samples from symptomatic patients with IBD in remission for proteomics, micro-RNA and microbial composition and to compare the results with findings in healthy participants and asymptomatic patients with IBD in remission.

Part 1 and 2. Anorectal manometry, barostat assessment and validated questionnaires in healthy volunteers and asymptomatic IBD patients.

Awareness of rectal filling is critical to normal bowel function. Abnormal visceral sensitivity and/or biomechanical function (most commonly described by evaluation of rectal compliance) is often found in fecal incontinence and evacuation disorders, providing the rationale for measurement of anorectal sensory and motor function.

Aims:

To determine the correlation between sensitivity testing and the level-of-agreement of rectal compliance testing between the HRAM and the barostat protocol.

To obtain normal values regarding anorectal function from healthy volunteers and asymptomatic IBD patients which will be used for comparison with the values obtained from symptomatic patients with IBD.

To obtain normal values regarding gastrointestinal symptoms and psychometric scales using standardized questionnaires, which will be used for comparison with the values obtained from symptomatic patients with IBD.

To obtain biological samples. Results of the analyses of these samples will be compared with the results from the symptomatic IBD patients as outlined in the part 6 of the research plan.

Design: reliability and method comparison study but at the same time the participants will constitute the control cases in the planed case control studies.

No data is available regarding normal values for rectal compliance using the HRAM method. In a study comparing a rapid non-elastic barostat bag measurement with a standardized barostat procedure, a total of 25 subjects was sufficient to detect a difference in sensitivity threshold volumes.

The following validated questionnaires will be used:

ROME IV diagnostic criteria, IBS symptom severity index, Gastrointestinal symptom severity scale, Bristol stool form scale, Nepean dyspepsia index, Depression Module (PHQ-9), Anxiety module (GAD-7), Symptomatic severity module (PHQ-15), Visceral sensitivity index, Assessment of disease-specific quality of life, Assessment of socioeconomic status of IBS patients, Assessment of personality (NEO-FFI-3), Vaizey score for incontinence.

HRAM The investigation consists of a series of pressure measurements that assess resting pressure of the anal canal, voluntary function during short and long squeeze, assessment of the cough reflex, rectoanal inhibitory reflex during rectal distension and rectoanal coordination and propulsive force during simulated defecation.

Rectal sensitivity testing and rectal compliance studies will be performed through inflation of an elastic balloon connected to the HRAM catheter, placed within the rectum. During inflation, perceived sensations are reported: first sensation, desire to defecate, urgency and maximum toleration or pain.

The distending volume and pressure will be recorded and the rectal compliance after correction for the internal compliance of the elastic balloon will be calculated (ΔV⁄ΔP).

Barostat protocol tests:

Ascending method of limits protocol: ramp inflation starting at 0 mmHg and increasing in steps of 4 mmHg for 1 min per step to a maximum of 60 mmHg. Thresholds for first sensation, first desire to defecate, urgency, discomfort and pain will be recorded and the rectal compliance calculated.

Random order phasic distensions protocol: phasic distensions (60 sec) of 12, 24, 36 and 48 mmHg above basic operating pressure (BOP) will be each applied once in a random order. The maximum pressure is limited by the pain threshold from the AML. The subjects will rate the intensity of four different sensations during the last 30 sec of each distension (gas, urgency, discomfort and pain).

Biological samples will be obtained during a separate visit to the gastroenterology department.

Part 3 and 4. Assessment of symptoms and anorectal function in patients with quiescent ulcerative colitis respective quiescent Crohns disease with anorectal involvement.

Aim To obtain values regarding anorectal function from patients with IBD in remission using the HRAM protocol and the standardized barostat protocol.

To phenotype the patients by obtaining data regarding gastrointestinal symptoms and psychometric values using standardized questionnaires, and to analyse these data together with the anorectal function data.

To obtain biological samples from symptomatic patients with IBD in remission

There are no data available regarding normal values for rectal compliance and sensitivity using the HRAM method in IBD patients. However, earlier studies, comparing healthy volunteers with IBS patients using a similar standardized barostat protocol, demonstrated that a total of 13 IBS patients and 13 healthy controls was sufficient to detect a difference in sensitivity threshold volumes and rectal compliance. For this reason, 15 patients will be included.

The same protocol as for part 1 will be applied.

Part 5. Assessment of IBS-like symptoms and psychological comorbidities in patients with UC and Crohn's disease in remission.

Increased visceral perception (hypersensitivity) with disturbed bidirectional brain-gut signaling is considered the biological hallmark of IBS.

Aim: to investigate whether patients with quiescent IBD meet the Rome IV criteria for IBS with concomitant psychological comorbidity, or that these patients suffer from gastrointestinal symptoms due to the effects of a long-lasting inflammatory process leading to rectal fibrosis. This knowledge has consequences for the treatment of these patients.

The HRAM measurements will be used to establish the presence of an eventual rectal motor dysfunction as the cause for symptoms. The barostat data will be used to establish whether there is a decreased rectal compliance, suggestive for fibrosis, as well as to establish whether the IBD patients show a visceral hypersensitivity, in comparison with healthy controls.

The symptom and psychometric questionnaires will be used to establish whether the quiescent IBD patients demonstrate a typical IBS phenotype with high comorbidities of anxiety, depression, somatization and a personality treat with a high level of neuroticism.

Part 6. Molecular profile of symptomatic patients with quiescent IBD compared to healthy volunteers and asymptomatic patients with quiescent IBD Aspects of gut microbiota, genome, transcriptome and proteome-profiles will be compared between the study groups.

The microbiological data will be combined with proteomic data from plasma and rectal biopsies, data from the mi-RNA analysis and correlated with data on the clinical and psychological phenotype of the patients. This "multi-omics" approach requires development of bioinformatics methods, which currently are underway in IBD studies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Symptomatic IBD patients: Moderate to severe IBD in remission with persistent symptoms as reported by symptom index and short health scale.
* Asymptomatic IBD patients: moderate to severe IBD in remission without symptoms

Exclusion Criteria:

Healthy volunteers:

* gastrointestinal disease, functional gastrointestinal symptoms,
* psychiatric disease
* anal or pelvic surgery, inclusive interventions during delivery
* diabetes, cardiovascular, renal, or hepatic disease,
* concurrent or recent treatment with drugs affecting intestinal function or mood (antidepressants), nutritional supplements or herb products affecting intestinal function (probiotics), abuse of alcohol or drugs, and a recent (< 2 weeks) history of systemic steroid therapy.

IBD patients

* active disease
* anal or pelvic surgery, inclusive interventions during delivery
* diabetes, cardiovascular, renal, or hepatic disease,
* concurrent or recent treatment with drugs affecting intestinal function or mood (antidepressants), nutritional supplements or herb products affecting intestinal function (probiotics), abuse of alcohol or drugs, and a recent (< 2 weeks) history of systemic steroid therapy. Patients taking antidiarrhoeal or laxatives can be included after a 48 h washout period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Remission is defined as endoscopic absence of active inflammation and f-calprotectin < 100 mg/kg.
  Moderate to severe disease is defined as patients treated with the immune modulating drugs thiopurine or methotrexate, and/or biological drugs infliximab, adalimumab, golimumab, vedolizumab or ustekinumab.
  Presence of symptoms is evaluated by the short health scale and symptom index questionnaires that all IBD patients fill before their visit to the outpatient ward.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Rectal compliance testing with the HRAM and Barostat methods | 15 minnutes
  RC is defined as the relation between volume (ml) respective pressure (mmHg) at half the maximum volume observed and at thresholds for first sensation, first urge, intense urge and maximum tolerated volume.
Rectal sensitivity testing with whit the HRAM and Barostat methods | 15 minutes
  RS is defined as the volume (ml) respective pressure (mmHg) observed at 4 (HRAM) respective 5 (Barostat) predefined sensation thresholds.
Anal squeeze pressure | 3 minutes
  Anal pressure in mmHg assessed from the best of three short squeezes (5seconds) and a prolonged squeeze of 30 seconds during the HRAM investigation.
Anal rest pressure | 3 minutes
  Anal rest pressure in mmHg assessed during the HRAM investigation.
Anorectal coordination during simulated defecation | 2 minutes
  Binary outcome. Anorectal coordination is assessed from the changes in rectal and anal pressure during simulated defecation. The outcomes are: Effective simulated defecation: yes/no
Dyssynergic defecation | 2 minutes
  Categorical binary outcome. Anorectal coordination is assessed from the changes in rectal and anal pressure during simulated defecation. The outcome is: dyssynergic defecation: yes/no
GI symptoms based on the GSRS-IBS questionaire | 10 minutes
  The answers are converted to a numerical value where the higher score corresponds to worse symptoms.
GI symptoms based on the IBS symptom severity index | 10 minutes
  The answers are converted to a numerical value where the higher score corresponds to worse symptoms.
GI specific anxiety based on the Visceral sensitivity index | 10 minutes
  The answers are converted to a numerical value where the higher score corresponds to worse symptoms.
Symptom severity based on the Symptomatic severity module (PHQ 12) | 10 minutes
  The answers are converted to a numerical value where the higher score corresponds to worse symptoms.
Assessment of personality using the NEO-FFI-3questionnaire (Big five inventory) | 20 minutes
  The NEO-FFI is a 44-item personality inventory that examines a person's Big Five personality traits (openness to experience, conscientiousness, extraversion, agreeableness, and neuroticism). Each item is assigned a value between 1 to 5 by the participant. Scores for each of the 5 personality traits are calculated and interpreted with the help of the adequate tables.
Pathogenic variants | 30 minutes
  Arrays such as Illumina Global Screening Array and available exonic content databases like ClinVar, will be used to define "Pathogenic" and "Likely Pathogenic" variants in the likelihood of developing a phenotype and the frequency of such alleles within a given population.
Genetical risk score. | 30 minutes
  The liability for the symptomatic phenotype will be calculated by the sum of an individual's risk alleles, weighted by risk allele effect sizes derived from genome-wide associated study data.
Methylation status | 30 minutes
  Commercially available arrays such as the Illumina infinium 450K methylation array will also be used for the analyses of methylation status.
Aspects of proteomics | 30 minutes
  Olink precision inflammatory panel allows simultaneous analysis of 92 inflammation-related protein biomarkers, both in serum and in the rectal mucosa. Thereafter, we will use the Ingenuity Pathway Analysis (IPA) which allows for matching the results of our data against earlier IPA analyses.
Aspects of microbiome. | 30 minutes
  Fecal microbiota as well as mucosa-associated microbiota will be analysed both for qualitative and quantitative composition with both 16S-RNA sequencing and next-generation metagenomic sequencing, to identify the bacterial profile in the patients.
Aspects of transcriptome | 30 minutes
  Blood samples (Pax-gene tubes) and Rectal biopsies will be used for extraction of miRNA and subsequent analysis. In order to analyze the total RNA expression, Next Generation Sequencing (NGS) will be used.
The correlation between proteomics in the mucosa and in blood | 30 minutes
  Olink® precision proteomics inflammatory panel which allows simultaneous analysis of 92 inflammation-related protein biomarkers, both in serum and in the rectal mucosa.

SECONDARY OUTCOMES:
Cough reflex during HRAM | 2 minutes
  Recto anal inhibitory reflex is defined as the drop in anal rest pressure observed after inflating a balloon in the rectum to 60 ml. The studies are interpreted as positive or negative and the amplitude of the pressure change is recorded.
RAIR reflex during HRAM | 2 minutes
  Cough reflex is the increase in anal pressure during cough. The studies are interpreted as positive or negative and the amplitude of the pressure change is recorded.
The adaptive function of the rectum during barostat investigation | 12 minutes
  The adaptive function of the rectum is defined as the change (increase) in volume necessary to maintain the same rectal pressure during the random phasic distensions of the barostat investigation.
The aggregate sensation intensity scores for gas | 12 minutes
  The visual analogue scale scores, in mm, marked by the patients at each distension during the random phasic distension part of the barostat study.
The aggregate sensation intensity scores for urgency | 12 minutes
  The visual analogue scale scores, in mm, marked by the patients at each distension during the random phasic distension part of the barostat study.
The aggregate sensation intensity scores for discomfort | 12 minutes
  The visual analogue scale scores, in mm, marked by the patients at each distension during the random phasic distension part of the barostat study.
The aggregate sensation intensity scores for pain | 12 minutes
  The visual analogue scale scores, in mm, marked by the patients at each distension during the random phasic distension part of the barostat study.
Stool consistence using the Bristol stool form scale | 10 minutes
  Categorical ordered variable assigning a numeric value to stool consistency. Higher values correspond to softer stools.
Dyspeptic symptoms using the Nepean dyspepsia index | 10 minutes
  The answers are converted to a numerical value where the higher score corresponds to worse symptoms.
Depression using the Depression Module (PHQ-9) | 15 minutes
  The answers are converted to a numerical value where the higher score corresponds to worse symptoms.
Aanxiety using the Anxiety module (GAD-7) | 15 minutes
  The answers are converted to a numerical value where the higher score corresponds to worse symptoms.
Assessment of disease-specific quality of life using the IBS-qol questionnaire | 15 minutes
  The answers are converted to a numerical value were the higher score corresponds to worse symptoms.
Incontinence using the Vaizey score for incontinence | 10 minutes
  The answers are converted to a numerical value where the higher score corresponds to worse symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Michiel van Nieuwenhoven, assoc prof, Principal Investigator — University Hospital Örebro
Locations (1):
- University hospital Örebro, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brochard C, Siproudhis L, Leveque J, Grouin A, Mallet AL, Bretagne JF, Ropert A, Bouguen G. Factors Associated with Fecal Incontinence in Women of Childbearing Age with Crohn's Disease. Inflamm Bowel Dis. 2017 May;23(5):775-780. doi: 10.1097/MIB.0000000000001056. PMID 28394805
- [Background] Kozeluhova J, Kotyza J, Balihar K, Krcma M, Cedikova M, Karbanova J, Kalis V, Janska E, Matejovic M. Risk of anal incontinence in women with inflammatory bowel diseases after delivery. Bratisl Lek Listy. 2017;118(6):328-333. doi: 10.4149/BLL_2017_072a. PMID 28664741
- [Background] Stewart DB Sr. Fecal Incontinence Among Patients With Crohn's Disease: Does Awareness Change Anything? Dis Colon Rectum. 2017 Aug;60(8):759-760. doi: 10.1097/DCR.0000000000000811. No abstract available. PMID 28682961
- [Background] Vollebregt PF, Visscher AP, van Bodegraven AA, Felt-Bersma RJF. Validation of Risk Factors for Fecal Incontinence in Patients With Crohn's Disease. Dis Colon Rectum. 2017 Aug;60(8):845-851. doi: 10.1097/DCR.0000000000000812. PMID 28682970
- [Background] Menees SB, Almario CV, Spiegel BMR, Chey WD. Prevalence of and Factors Associated With Fecal Incontinence: Results From a Population-Based Survey. Gastroenterology. 2018 May;154(6):1672-1681.e3. doi: 10.1053/j.gastro.2018.01.062. Epub 2018 Feb 3. PMID 29408460
- [Background] Simren M, Axelsson J, Gillberg R, Abrahamsson H, Svedlund J, Bjornsson ES. Quality of life in inflammatory bowel disease in remission: the impact of IBS-like symptoms and associated psychological factors. Am J Gastroenterol. 2002 Feb;97(2):389-96. doi: 10.1111/j.1572-0241.2002.05475.x. PMID 11866278
- [Background] Minderhoud IM, Oldenburg B, Wismeijer JA, van Berge Henegouwen GP, Smout AJ. IBS-like symptoms in patients with inflammatory bowel disease in remission; relationships with quality of life and coping behavior. Dig Dis Sci. 2004 Mar;49(3):469-74. doi: 10.1023/b:ddas.0000020506.84248.f9. PMID 15139501
- [Background] Bondurri A, Maffioli A, Danelli P. Pelvic floor dysfunction in inflammatory bowel disease. Minerva Gastroenterol Dietol. 2015 Dec;61(4):249-59. Epub 2015 Nov 23. PMID 26603727
- [Background] Fukuba N, Ishihara S, Tada Y, Oshima N, Moriyama I, Yuki T, Kawashima K, Kushiyama Y, Fujishiro H, Kinoshita Y. Prevalence of irritable bowel syndrome-like symptoms in ulcerative colitis patients with clinical and endoscopic evidence of remission: prospective multicenter study. Scand J Gastroenterol. 2014 Jun;49(6):674-80. doi: 10.3109/00365521.2014.898084. Epub 2014 Mar 20. PMID 24646420
- [Background] Ansari R, Attari F, Razjouyan H, Etemadi A, Amjadi H, Merat S, Malekzadeh R. Ulcerative colitis and irritable bowel syndrome: relationships with quality of life. Eur J Gastroenterol Hepatol. 2008 Jan;20(1):46-50. doi: 10.1097/MEG.0b013e3282f16a62. PMID 18090990
- [Background] Halpin SJ, Ford AC. Prevalence of symptoms meeting criteria for irritable bowel syndrome in inflammatory bowel disease: systematic review and meta-analysis. Am J Gastroenterol. 2012 Oct;107(10):1474-82. doi: 10.1038/ajg.2012.260. Epub 2012 Aug 28. PMID 22929759
- [Background] Spiller R, Lam C. The shifting interface between IBS and IBD. Curr Opin Pharmacol. 2011 Dec;11(6):586-92. doi: 10.1016/j.coph.2011.09.009. Epub 2011 Oct 13. PMID 22000604
- [Background] Carrington EV, Scott SM, Bharucha A, Mion F, Remes-Troche JM, Malcolm A, Heinrich H, Fox M, Rao SS; International Anorectal Physiology Working Group and the International Working Group for Disorders of Gastrointestinal Motility and Function. Expert consensus document: Advances in the evaluation of anorectal function. Nat Rev Gastroenterol Hepatol. 2018 May;15(5):309-323. doi: 10.1038/nrgastro.2018.27. Epub 2018 Apr 11. PMID 29636555
- [Background] Loening-Baucke V, Metcalf AM, Shirazi S. Anorectal manometry in active and quiescent ulcerative colitis. Am J Gastroenterol. 1989 Aug;84(8):892-7. PMID 2756980
- [Background] Brochard C, Siproudhis L, Ropert A, Mallak A, Bretagne JF, Bouguen G. Anorectal dysfunction in patients with ulcerative colitis: impaired adaptation or enhanced perception? Neurogastroenterol Motil. 2015 Jul;27(7):1032-7. doi: 10.1111/nmo.12580. Epub 2015 May 4. PMID 25940976
- [Background] Chen P, Zhou G, Lin J, Li L, Zeng Z, Chen M, Zhang S. Serum Biomarkers for Inflammatory Bowel Disease. Front Med (Lausanne). 2020 Apr 22;7:123. doi: 10.3389/fmed.2020.00123. eCollection 2020. PMID 32391365
- [Background] D'Haens G, Rieder F, Feagan BG, Higgins PDR, Panes J, Maaser C, Rogler G, Lowenberg M, van der Voort R, Pinzani M, Peyrin-Biroulet L, Danese S; International Organization for Inflammatory Bowel Disease Fibrosis Working Group. Challenges in the Pathophysiology, Diagnosis, and Management of Intestinal Fibrosis in Inflammatory Bowel Disease. Gastroenterology. 2022 Jan;162(1):26-31. doi: 10.1053/j.gastro.2019.05.072. Epub 2019 Jun 27. PMID 31254502
- [Background] Vanhoutvin SA, Troost FJ, Kilkens TO, Lindsey PJ, Jonkers DM, Venema K, Masclee A, Brummer RJ. Alternative procedure to shorten rectal barostat procedure for the assessment of rectal compliance and visceral perception: a feasibility study. J Gastroenterol. 2012 Aug;47(8):896-903. doi: 10.1007/s00535-012-0543-x. Epub 2012 Feb 24. PMID 22361864
- [Background] Mavroudis G, Strid H, Jonefjall B, Simren M. Visceral hypersensitivity is together with psychological distress and female gender associated with severity of IBS-like symptoms in quiescent ulcerative colitis. Neurogastroenterol Motil. 2021 Mar;33(3):e13998. doi: 10.1111/nmo.13998. Epub 2020 Oct 9. PMID 33034406
- [Background] Spiller RC, Humes DJ, Campbell E, Hastings M, Neal KR, Dukes GE, Whorwell PJ. The Patient Health Questionnaire 12 Somatic Symptom scale as a predictor of symptom severity and consulting behaviour in patients with irritable bowel syndrome and symptomatic diverticular disease. Aliment Pharmacol Ther. 2010 Sep;32(6):811-20. doi: 10.1111/j.1365-2036.2010.04402.x. PMID 20629976
- [Background] Halfvarson J, Brislawn CJ, Lamendella R, Vazquez-Baeza Y, Walters WA, Bramer LM, D'Amato M, Bonfiglio F, McDonald D, Gonzalez A, McClure EE, Dunklebarger MF, Knight R, Jansson JK. Dynamics of the human gut microbiome in inflammatory bowel disease. Nat Microbiol. 2017 Feb 13;2:17004. doi: 10.1038/nmicrobiol.2017.4. PMID 28191884
- [Background] Carstens A, Roos A, Andreasson A, Magnuson A, Agreus L, Halfvarson J, Engstrand L. Differential clustering of fecal and mucosa-associated microbiota in 'healthy' individuals. J Dig Dis. 2018 Dec;19(12):745-752. doi: 10.1111/1751-2980.12688. PMID 30467977
- [Background] Andersson E, Bergemalm D, Kruse R, Neumann G, D'Amato M, Repsilber D, Halfvarson J. Subphenotypes of inflammatory bowel disease are characterized by specific serum protein profiles. PLoS One. 2017 Oct 5;12(10):e0186142. doi: 10.1371/journal.pone.0186142. eCollection 2017. PMID 28982144